CLINICAL TRIAL: NCT04817566
Title: Neuromodulation Through Brain Stimulation-assisted Cognitive Training in Patients With Post-chemotherapy Cognitive Impairment
Brief Title: Cognitive Training and Brain Stimulation in Women With Post-chemotherapy Cognitive Impairment
Acronym: NeuroMod-PCCI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medicine Greifswald (Other)
Collaborators: University of Greifswald (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NeuroMod-PCCI
Record Dates: First submitted 2021-03-24; First posted 2021-03-26 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer; Cognitive Impairment
MeSH Terms: conditions — Breast Neoplasms; Cognitive Dysfunction | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- stimulation group (Experimental): Anodal tDCS+ intensive cognitive Training
  Interventions: Device: Anodal tDCS; Behavioral: Intensive cognitive training
- sham group (Sham Comparator): Sham tDCS + intensive cognitive Training
  Interventions: Device: Sham tDCS; Behavioral: Intensive cognitive training

INTERVENTIONS:
Device: Anodal tDCS — Anodal transcranial direct current stimulation (tDCS), 9 sessions with 20 minutes stimulation each (2 mA).
  Arms: stimulation group
Device: Sham tDCS — Sham transcranial direct current stimulation (tDCS), 9 sessions with 30 sec stimulation each (2 mA) to ensure blinding of participants.
  Arms: sham group
Behavioral: Intensive cognitive training — Intensive cognitive training of a letter memory updating task, 9 sessions for approximately 20 min

SUMMARY:
The aim of this study is to investigate whether a high definition tDCS-accompanied intensive cognitive training of working memory leads to performance improvement in women with post-chemotherapy cognitive impairment after breast cancer treatment.

DETAILED DESCRIPTION:
Patients who have undergone chemotherapy, may develop post-chemotherapy cognitive impairment (PCCI), which may occur in several cognitive domains and persist for many years. These declines in cognitive functions can lead to psychological distress and affect overall patients' quality of life. The goal of the present study is to assess behavioral effects of a multi-session cognitive training combined with high-definition transcranial direct current stimulation (tDCS) in women with PCCI. First studies have shown positive effects of cognitive training on trained and untrained functions and the subjective perception of stress, however the effects are small and transfer effects are inconsistent. A promising approach to elongate and increase the effects of cognitive training is to combine the training with tDCS. Therefore, in this study women with PCCI will participate in a three-week cognitive training with concurrent online high-definition tDCS application. Cognitive performance (primary), as well as Quality of Life scores and Sleep data will be examined before, during and after the intervention. In order to draw conclusions about the effect of tDCS in addition to cognitive training, a control group, receiving sham stimulation during training, will be assessed. A Follow-up session to assess long-term effects is planned four weeks after the post assessment. The results of the study will offer valuable insights into efficacy of combined tDCS and cognitive training intervention in women with PCCI in order to establish its potential to induce improvements in cognitive functions, and to beneficially affect patient-reported outcome measures.

ELIGIBILITY:
Inclusion Criteria:

1. Chemotherapy to treat breast cancer (≥ 6 months post-treatment).
2. Self-reported concerns regarding cognitive functioning.
3. Age: 18-65 years.
4. right-handedness

Exclusion Criteria:

1. History of dementia before treatment of cancer.
2. Other neurodegenerative neurological disorders; epilepsy or history of seizures.
3. Severe and untreated medical conditions that preclude participation in the training, as determined by responsible physician.
4. History of moderate to severe substance use disorder according to DSM-5
5. Moderate to severe acute psychiatric disorders according to DSM-5
6. Contraindication to tDCS application (Antal et al., 2017)

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2021-11-02 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Working memory performance at post-assessment | 3 weeks
  Performance in a near transfer task (n-back) under anodal tDCS compared to sham condition; operationalized by % correct responses in the n-back task

SECONDARY OUTCOMES:
Working memory performance at follow-up assessment | 4 weeks after training
  Performance in a near transfer task (n-back) under anodal tDCS compared to sham condition; operationalized by % correct responses in the n-back task
Working memory training performance (Letter Updating Task) at post-assessment | 3 weeks
  Performance in primary memory training task (Letter Updating Task) at post-assessment, operationalized by number of correctly recalled lists in the letter updating task
Working memory training performance (Letter Updating Task) at follow-up assessment | 4 weeks after training
  Performance in primary memory training task (Letter Updating Task) at follow-up assessment, operationalized by number of correctly recalled lists in the letter updating task
Quality of Life at post-assessment | 3 weeks
  PROMIS score for HRQoL (PROPr score) and scores of subscales (e.g. cognitive function)
Quality of Life at follow-up assessment | 4 weeks after training
  PROMIS score for HRQoL (PROPr score) and scores of subscales (e.g. cognitive function)
Visuo-spatial performance at post-assessment | 3 weeks
  Visuo-spatial performance at post-assessment operationalized by number of correctly recalled items in the VR task.
Visuo-spatial performance at follow-up assessment | 3 weeks
  Visuo-spatial performance at follow-up assessment operationalized by number of correctly recalled items in the VR task.

CONTACTS AND LOCATIONS:
Overall Officials: Agnes Flöel, Prof., Study Director — University Medicine Greifswald
Locations (1):
- University Medicine Greifswald, Greifswald, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Rocke M, Knochenhauer E, Thams F, Antonenko D, Fromm AE, Jansen N, Aziziaram S, Grittner U, Schmidt S, Vogelgesang A, Brakemeier EL, Floel A. Neuromodulation through brain stimulation-assisted cognitive training in patients with post-chemotherapy subjective cognitive impairment (Neuromod-PCSCI) after breast cancer: study protocol for a double-blinded randomised controlled trial. BMJ Open. 2025 May 21;15(5):e096162. doi: 10.1136/bmjopen-2024-096162. PMID 40398955